CLINICAL TRIAL: NCT01292148
Title: Core Temperature Measurement in Therapeutic Hypothermia: Tympanic Membrane, Bladder and Rectal Versus Pulmonary Artery Methods
Brief Title: Measurement of Core Temperatures During Therapeutic Hypothermia
Acronym: TH
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Shin, Seoul National University, Seoul National University Hospital
Other Study IDs: MCT-TH
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Arrest
Keywords: resuscitation, hypothermia
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine that the measurements of rectal and bladder temperature are correctly consistent with core temperature by using the pulmonary artery catheter during therapeutic hypothermia; rapid cooling, maintenance, and slow rewarming phase.

DETAILED DESCRIPTION:
The guidelines of therapeutic hypothermia(TH)are rapid cooling, from normothermia to mild hypothermia(32~34 degree), maintenance, and slow rewarming phase. If core temperature maintained below 32 degree during TH, som complications will be developed, such as arrythmia, hypotension, cold diuresis, coagulopathy, and so on. Therefore correct measurement of core temperature during TH is very important process for successful post cardiac arrest care. we will know that rectal or bladder temperature are really reflect the core temperature during TH for post cardiac arrest care, especially rapid cooling phase, maintenance phase, and slow rewarming phase, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Out of cardiac arrest patient who is 18 years old.
* Mean arterial pressure must be over 65 mmHg after return of spontaneous circulation.
* Family consent to this study.

Exclusion Criteria:

* In hospital arrest.
* Arrest due to trauma
* Arrest due to intracranial hemorrhage.
* Below 30 degree at initial core temperature.
* Pregnancy.
* Family do not agree with our study.
* Active bleeding patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post cardiac arrest care with therapeutic hypothermia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference of core temperature between rectum, bladder, esophagus and pulmonary artery | During 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Shin JongHwan, Principal Investigator — Seoul National University Boramae Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, South Korea